CLINICAL TRIAL: NCT07124351
Title: Intraoperative Imaging of Gastrointestinal Malignancies Using Pafolacianine (CYTALUX™)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: On Target Laboratories, LLC (Industry)
Responsible Party: Principal Investigator, Miguel Burch, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00003515
Record Dates: First submitted 2025-07-31; First posted 2025-08-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Gastrointestinal Cancer; Gastric Cancer; Esophageal Cancer; Appendiceal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Appendiceal Neoplasms | interventions — Pafolacianine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- CYTALUX™ (pafolacianine) (Experimental): Enrolled subjects will be dosed with 0.025 mg/kg CYTALUX™ (pafolacianine) injection intravenously, with the hour-long infusion completing from 1 hour to up to 24 hours prior to imaging for the planned surgery.
  Interventions: Drug: CYTALUX™ (pafolacianine)

INTERVENTIONS:
Drug: CYTALUX™ (pafolacianine) — All subjects participating in the study are expected to receive CYTALUX™ (pafolacianine) injection and standard care surgery; 1 to 24 hours after CYTALUX™ (pafolacianine) injection infusion is completed, all tumors planned to be removed as part of standard care will undergo assessment with NIR light imaging both intraoperatively and on the back table following surgery.

SUMMARY:
This is an open-label study in adults to determine feasibility of using CYTALUX™ (pafolacianine) injection with near-infrared (NIR) fluorescent imaging for detecting any type adenocarcinoma (gastric, esophageal and appendiceal).

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age and older of any sex.
2. Have a primary diagnosis, or a high clinical suspicion, of gastroesophageal adenocarcinoma based on CT (computed tomography)/PET (positron emission tomography) or other imaging (Cohort 1) or diagnosis of appendiceal adenocarcinoma with a high clinical suspicion of peritoneal carcinomatosis (Cohort 2).
3. Have an indication for surgical intervention for gastroesophageal tumor resection or diagnostic laparoscopy for assessment of peritoneal disease burden.
4. Willingness to stop the use of folate, folic acid, or folate-containing supplements within 48 hours before administration of CYTALUX.
5. Willingness of research participant to give written informed consent.

Exclusion Criteria:

1. Any medical condition that in the opinion of the investigators could potentially jeopardize the safety of the subject.
2. History of anaphylactic reactions to products containing indocyanine green for near infrared imaging. Subjects with a medical history of 'idiopathic anaphylaxis' will require evaluation.
3. History of allergy to any of the components of CYTALUX™ (pafolacianine) injection.
4. Presence of any psychological, familial, sociological condition or geographical challenges potentially hampering compliance with the study protocol or follow-up schedule.
5. Known sensitivity to fluorescent light.
6. Women of childbearing potential who are pregnant or plan to become pregnant during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility of CYTALUX™ (pafolacianine) with near-infrared (NIR) fluorescent imaging | 12 months
  Determine feasibility of using CYTALUX™ (pafolacianine) injection with near-infrared (NIR) fluorescent imaging for detecting any type adenocarcinoma (gastric, esophageal and appendiceal) in at least 70% of the patients.

SECONDARY OUTCOMES:
Number of Lesions | 12 months
  Number of lesions that are simultaneously fluorescence positive and cancer positive.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Burch, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States